CLINICAL TRIAL: NCT00492466
Title: A Multicentre, Open Label, Non-Comparative Trial Investigating the Recovering of INF-Beta Efficacy in Breakthrough Relapsing-Remitting Multiple Sclerosis Patients With Neutralizing Interferon-Beta Antibodies
Brief Title: Investigating if Interferon-Beta Can be Used in Patients With MS After They Have Developed Neutralizing Antibodies
Acronym: RECOVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: biogen Idec MD, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECOVER
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; antibody; Neutralizing antibody; Binding antibody; MxA protein
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Interferon-beta-1a; Drug: methylprednisolone

INTERVENTIONS:
Drug: Interferon-beta-1a — dosage and frequency as per label
  Other Names: Avonex
Drug: methylprednisolone — dosage and frequency as per Biogen Idec protocol

SUMMARY:
This study is to find out if Interferon-beta can recover its effectiveness in patients with Multiple Sclerosis who have previously developed neutralizing antibodies to Interferon-Beta.

DETAILED DESCRIPTION:
This is a multi-center, open Label, non-comparative Phase IV trial. Eligible Patients will receive treatment with Interferon-beta-1a (AVONEX) 30mcg I.M. once weekly for up to 12 months.

In the wash-out period prior to commencing treatment with AVONEX, patients will receive treatment with intermittent Methylprednisolone 500 mg PO Daily for three consecutive days at monthly intervals.

The patients will be examined clinically and laboratory tests will be performed at screening (month -1) and after 3, 9, and 15 months.

Neutralizing antibody(NAb)titres and Binding antibody(BAb)titres as well as MxA protein levels will be evaluated at screening/baseline (month -1/0) and after 3, 6, 9, 12, and 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting Multiple Sclerosis according to Poser criteria (CDMS or LDMS) or Multiple Sclerosis according to McDonald criteria
* Disability equivalent to EDSS of 6.0 or less
* Clinical activity defined as at least one relapse rate within the last 12 months
* NAb titre >20 (measured at least 48 hours after last interferon-beta injection
* has been treated with subcutaneously administered interferon-beta-1b or interferon-beta-1a (Rebif) for at least 24 hours before enrollment

Exclusion Criteria:

* Any condition that might give rise to similar symptoms as MS
* Immunomodulatory therapy other than interferon-beta-1a or interferon-beta-1b or any immunosuppressive treatment six months prior to inclusion into the trial
* Treatment with glucocorticoids or ACTH less than one month prior to inclusion into the trial
* History of major depression
* Alcohol or drug dependency
* Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV)
* hypertension (BP > 180/110 mmHg)
* Renal insufficiency defined as serum creatinine > 1.5 times the upper normal reference limit
* Any systemic disease that can influence the patient's safety and compliance, or the evaluation of the disability
* Gastro-intestinal ulcers, gastritis, or dyspepsia
* Women who are pregnant, breast-feeding or have the possibility for pregnancy during the trial. To avoid pregnancy, women have to be postmenopausal, surgical sterile, sexually inactive or practice reliable contraceptives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Reduction in the proportion of patients being neutralizing antibody (NAb) positive (titre>20) | Month -1 and after 3, 6, 9, 12, and 15 months

SECONDARY OUTCOMES:
Change in MxA protein values | Month -1 and after 3, 6, 9, 12, and 15 months
Change in binding antibody (Bab) tires | Month -1 and after 3, 6, 9, 12, and 15 months
Proportion of patients with NAb positive titre <5 | Month -1 and after 3, 6, 9, 12, and 15 months
Change in annualised relapse rate | at 3, 6, 9, 12, and 15 months
The number of relapse-free patients | at 3, 6, 9, 12, and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — neurologyclinicaltrials@biogenidec.com
Locations (1):
- Coordinating Research Site, Turku, Finland